CLINICAL TRIAL: NCT00442455
Title: Phase I/II Trial of Erlotinib, Radiation Therapy, and Cisplatin in Patients With Complete Resected Squamous Cell Carcinoma of the Head and Neck
Brief Title: Erlotinib,Radiation and Cisplatin in Patients With Complete Resected Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Responsible Party: Principal Investigator, Lola, Oncologist, Grupo de Investigación Clínica en Oncología Radioterapia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML 18729
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-05

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Head Neck Carcinoma Erlotinib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib, radiotherapy. (Experimental): There are three cohorts of patients in whom the dose of Erlotinib chlorhydrate(100 and 150 mg) and Cisplatin (30 and 40 mg / m2) will be increase, and the doses of Radiation therapy being fixed (63 Gy during 5 days a week during 7 weeks)
  Interventions: Drug: Erlotinib chlorhydrate; Drug: Cisplatin; Procedure: Radiation therapy

INTERVENTIONS:
Drug: Erlotinib chlorhydrate — 150 mg/day for 7 weeks
  Other Names: Erlotinib clorhidrate
Drug: Cisplatin — 30 mg/m2 i.v. weekly for 7 weeks
  Other Names: Cisplatino
Procedure: Radiation therapy — 63 Gy, five days a week, for 7 weeks

SUMMARY:
The purpose of the study is to determinate the free-progression interval in patients with surgically resected locally advanced squamous cell carcinoma of head and neck treated with the maximum tolerated dose of the combination of erlotinib, radiation therapy and cisplatin, previously established in a safety trial.

DETAILED DESCRIPTION:
Phase I:

3 cohorts of 3-6 patients, patients will received:

* Erlotinib 100-150 mg/day po for 7 weeks.
* Cisplatin 30-40 mg/m2 iv weekly for 7 weeks.
* Radiation therapy 63 Gy, five days a week, for 7 weeks. Cohort 1: 3 patients will be included in cohort 1.

If no DLT has been recorded in the first three patients during the 7-weeks treatment, the dose level of erlotinib will be escalated to 150 mg and enrollment of cohort 2 will be initiated.

If DLT has been recorded in one out of the first three patients during the during the 7-weeks treatment, then the first cohort will be expanded to 6 patients.

* If no further DLT has been recorded in patients 4 to 6 of cohort 1 during the 7-weeks treatment cycle, the dose level of erlotinib will be escalated to 150 mg and enrollment of cohort 2 will be initiated, after patient 6 has completed the 7-weeks treatment.
* If DLT has been recorded in one out of the patients 4 to 6 of cohort 1 during the 7-weeks treatment cycle, the dose level of erlotinib will be escalated to 150 mg and enrollment of cohort 2 will be initiated, after patient 6 has completed the 7-weeks treatment.
* If DLT has been recorded in 2 patients of the patients 4 to 6 of cohort 1, during the during the 7-weeks treatment, then the trial will be terminated and this dose level will be considered as the Maximum Tolerated Dose (MTD).

If DLT has been recorded in 2 patients of the first three patients during the during the 7-weeks treatment, then the trial will be terminated and this dose level will be considered as the Maximum Tolerated Dose (MTD).

Cohort 2:

If DLT has been recorded in one out of the first three patients or 1-2 of the 6 patients in cohort 1, 3 patients will be included in cohort 2.

If no DLT has been recorded in the first three patients during the 7-weeks treatment, the dose level of cisplatin will be escalated to 40 mg/m2 and enrollment of cohort 3 will be initiated.

If DLT has been recorded in one out of the first three patients during the during the 7-weeks treatment, then the second cohort will be expanded to 6 patients.

* If no further DLT has been recorded in patients 4 to 6 of cohort 2 during the 7-weeks treatment cycle, the dose level of cisplatin will be escalated to 40 mg/m2 and enrollment of cohort 3 will be initiated, after patient 6 has completed the 7-weeks treatment
* If DLT has been recorded in one out of the patients 4 to 6 of cohort 2 during the 7-weeks treatment cycle, the dose level of cisplatin will be escalated to 40 mg/m2 and enrollment of cohort 3 will be initiated, after patient 6 has completed the 7-weeks treatment
* If DLT has been recorded in 2 patients of the patients 4 to 6 of cohort 2 during the during the 7-weeks treatment, then the trial will be terminated and this dose level will be considered as the Maximum Tolerated Dose (MTD).

If DLT has been recorded in 2 patients of the first three patients of cohort 2 during the during the 7-weeks treatment, then the trial will be terminated and this dose level will be considered as the Maximum Tolerated Dose (MTD).

Cohort 3:

If DLT has been recorded in one out of the first three patients or 1-2 of the 6 patients in cohort 2, 3 patients will be included in cohort 2.

If no DLT has been recorded in the first three patients during the 7-weeks treatment, then the Maximum Tolerated Dose has not been reached.

If DLT has been recorded in one out of the first three patients during the during the 7-weeks treatment, then the third cohort will be expanded to 6 patients.

* If no further DLT has been recorded in patients 4 to 6 of cohort 3 during the 7-weeks treatment cycle, then the Maximum Tolerated Dose has not been reached.
* If DLT has been recorded in one out of the patients 4 to 6 of cohort 3 during the 7-weeks treatment cycle, then the Maximum Tolerated Dose has not been reached.
* If DLT has been recorded in 2 patients of the patients 4 to 6 of cohort 3 during the during the 7-weeks treatment, then the trial will be terminated and this dose level will be considered as the Maximum Tolerated Dose (MTD).

If DLT has been recorded in 2 patients of the first three patients of cohort 3 during the during the 7-weeks treatment, then the trial will be terminated and this dose level will be considered as the Maximum Tolerated Dose (MTD).

Inclusion of the third patient of each cohort will not be allowed until the safety data from the two previous patients have been analyzed

Inclusion of the third patient of each cohort will not be allowed until the safety data from the two previous patients have been analyzed

DLT is defined as:

* Any clinically intolerable hematological or non-hematological grade 3-4 toxicity.
* Grade 3-4 diarrhoea.
* Grade 3-4 or clinically intolerable grade 2 skin rash.
* Grade 4 mucositis implying a temporary interruption of radiation therapy (for longer than 2 consecutive weeks).
* Grade 4 mucositis occurring within the first 3 weeks of treatment.
* Grade 3-4 mucositis accompanied by one of the following toxicities:
* Worsening of performance status, defined as ECOG ≥ 2 or a decrease of 40% in the Karnofsky performance status scale.
* Grade 3 Weight loss (corresponding to a weight loss of ≥ 20% with respect to baseline weight).
* Underlying pain (not including swallowing) VAS > 7.
* Parenteral nutrition.
* Any clinically significant toxicity, involving treatment interruption for a period longer than two weeks.

Maximum Tolerated Dose is defined as the dose level at which 2 patients of the first three patients of one cohort or ≥ 3 of the 6 patients of one cohort exhibit one DLT, during the 7-weeks treatment.

Phase II:

75 patients will be treated at dose step below MTD to determinate:

* Progression Free Survival, defined as the period of time from the surgery until disease progression or death.
* Overall survival.
* Locoregional progression-free survival.

A tumor assessment will be performed 30 days after the end of treatment and every 3 months until disease progression afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proof of epidermoid carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx, treated with surgical resection with curative intent.
* Surgical resection must have taken place within 8 weeks prior to the patient's inclusion in the study.
* In those patients having clinical regional lymph node involvement radical neck dissection is mandatory. However, radical neck dissection is not an inclusion criterion in patients staged as N0.
* Age 18-70 years.
* Anticipated life expectancy of ≥ 12 weeks.
* Patients should have at least one of the following criteria:

  1. Pathological T3-4 tumor stage, apart from T3N0 of the larynx with negative margins
  2. Pathological N2-3 nodal stage.
  3. Unfavorable pathological findings such as extranodal spread, positive resection margins, perineural and/or vascular involvement.
* Written informed consent given by the patient.
* Therapeutic compliance of the patient and geographical proximity to the hospital to facilitate appropriate follow-up.
* ECOG 0-1.
* No distant metastatic disease.
* Adequate organ function according to the following criteria:

  1. Adequate bone marrow reserve: ANC > 1,5 x 10(9) cells/L; Platelet count > 100 x 10(9) cells/L; Hemoglobin > 9 g/dL
  2. Liver function: Bilirubin < 1.5 x ULN; Alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0 x ULN
  3. Renal function: calculated creatinine clearance (CrCl) > 60ml/min or Creatinine (Cr) < 1.5 ULN of the reference laboratory.
  4. Serum calcium and alkaline phosphatase must be normal.
* Women of child bearing potential must have a negative pregnancy test within the 48h prior to the start of the treatment.
* Patients of both genders at a fertile age must follow effective contraceptive measures.
* Absence of symptomatic coronary artery disease or acute myocardial infarction within 6 months prior to study.
* Patients capable of oral deglutition or requiring gastrostomy.
* No problems of intestinal transit such as malabsorption syndrome, chronic inflammatory bowel disease and other diseases, which might impair drug absorption

Exclusion Criteria:

* Histology other than squamous cell carcinoma.
* Presence of macroscopic residual disease.
* Previous treatment with chemotherapy or radiotherapy or EGFR-targeted agents.
* Incomplete resection of the primary tumor or incomplete neck dissection.
* Patients being diagnosed with any other malignant disease, excluding resected nonmelanoma skin cancer or resected uterine cervix carcinoma.
* Pregnant or nursing women.
* Active infection.
* Concomitant severe illness (according to the opinion of the investigator) or whose estimated survival for this concomitant pathology is lower than that estimated for the neoplasm disease.
* Uncontrolled psychiatric illness.
* Inability to take oral medication, requiring intravenous feeding or prior surgical procedures affecting absorption or having active peptic ulcer.
* Impossibility to appropriate follow-up.
* Evidence of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding suggesting a condition that contraindicates the use of the study medication (erlotinib, cisplatin, radiotherapy), which might interfere with the analysis of the results or increase the risk of treatment complications.
* Any known significant ophthalmologic abnormalities, including severe xerophthalmia, keratoconjunctivitis sicca, Sjögren syndrome, severe exposure keratopathy or other abnormalities, which may increase the risk of corneal epithelial damage (the use of contact lenses during the study may increase the risk of corneal damage and its use is strongly discouraged. Those patients still using contact lenses will need a closer ophthalmologic follow-up.
* Frequent vomiting or medical disorder impairing swallowing of drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Determinate the maximum tolerated dose (PHASE I) | 17/MAR/08
Progression free survival (PHASE II) | 5 years

SECONDARY OUTCOMES:
DLT (PHASE I) | 17/MAR/08
Overall survival and locoregional progression free survival (PHASE II) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Calvo Manuel, Dr., Study Director — Hospital General Universitario Gregorio Marañón; Alejandro de la Torre Tomás, Dr., Principal Investigator — Hospital Universitario Clínica Puerta de Hierro; Manuel de las Heras González, Dr., Principal Investigator — Hospital San Carlos, Madrid; Ismael Herruzo Cabrera, Dr., Principal Investigator — Hospital Regional Universitario Carlos Haya; Fernando Arias de la Vega, Dr., Principal Investigator — Hospital de Navarra
Locations (5):
- Spain (5):
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Clínica Puerta de Hierro, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga